CLINICAL TRIAL: NCT01174992
Title: A Randomized, Controlled Study to Evaluate the Safety and Effectiveness of EVICEL as an Adjunct to Sutured Dural Repair
Brief Title: A Study to Evaluate the Safety and Effectiveness of EVICEL as an Adjunct to Sutured Dural Repair
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Collaborators: OMRIX Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 400-09-001; 2009-016501-41 (EudraCT Number)
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Dura Defects
Keywords: Fibrin sealant; CSF leak
MeSH Terms: conditions — Cerebrospinal Fluid Otorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evicel (Experimental)
  Interventions: Biological: Evicel
- Sutures only (Other)
  Interventions: Other: Sutures only

INTERVENTIONS:
Biological: Evicel — EVICEL is a human plasma derived fibrin sealant
  Arms: Evicel
Other: Sutures only — Standard of care
  Arms: Sutures only

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of EVICEL for use as an adjunct to dura sutures in elective cranial surgery to provide intraoperative watertight closure.

DETAILED DESCRIPTION:
This is a randomized, multi-center controlled study evaluating the effectiveness of EVICEL* as an adjunct to sutured dural closure compared to control to obtain an intraoperative watertight dural closure.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective craniotomy/craniectomy
* Age greater than or equal to 18 years
* Patients who are able and willing to comply with the procedures required by the protocol.
* Signed and dated written informed consent from the subject or from his/her legal representative prior to any study-related procedures.

Exclusion Criteria:

* Chemotherapy or radiation therapy within 7 days following surgery.
* Conditions compromising the immune system.
* Known hypersensitivity to the components (human fibrinogen, arginine hydrochloride, glycine, sodium chloride, sodium citrate, calcium chloride, human thrombin, human albumin, mannitol and sodium acetate) of the investigational product.
* Female subjects of childbearing potential with a positive pregnancy test prior to surgery.
* Female subjects who are breastfeeding or intend to become pregnant during the clinical study period.
* Participation in another clinical trial with exposure to another investigational drug or device within 30 days prior to enrollment.
* Major intraoperative findings or complications identified by the surgeon that may preclude conduct of the planned surgical procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Proportion of success | Day 1 (intraoperative)
  Proportion of success (intraoperative watertight closure) in the treatment of intraoperative CSF leakage.

SECONDARY OUTCOMES:
Incidence of CSF leakage | Day 5 post-op
Incidence of CSF leakage | Day 30 post-op
Incidence of adverse events | up to 30 days post-op
Incidence of surgical site infections | Day 5 and 30 post-op

CONTACTS AND LOCATIONS:
Overall Officials: James Hart, MD, Study Director — Ethicon, Inc.
Locations (12):
- Belgium (2):
  - Department of Neurosurgery, Ziekenhuis Oost Limburg, Genk
  - Department of Neurosurgery, University Hospital of Liège, Liège
- Department of Neurosciences and Rehabilitation, Tampere University Hospital, Tampere, Finland
- Service de Neurochirurgie B, Hopital Neurologique de Lyon, Cedex, France
- Germany (4):
  - Klinik für Neurochirurgie, Universitätsklinikum Essen, Essen
  - Department of Neurosurgery, University Giessen-Marburg, Giessen
  - Department of Neurosurgery, Klinikum Ingolstadt GmbH, Ingolstadt
  - Department of Neurosurgery University Clinics of Schleswig-Holstein Campus Kiel, Kiel
- VU Medical Centre, Amsterdam, Netherlands
- United Kingdom (3):
  - Department of Neurosurgery, John Radcliffe Hospital, Headington, Oxford
  - Department of Neurosurgery, Ninewells Hospital & Medical School, Dundee
  - Edinburgh Centre for Neuro-Oncology, Western General Hospital, Edinburgh